CLINICAL TRIAL: NCT00076830
Title: Investigations of Bone-Related Connective Tissue Disorders
Brief Title: Evaluation and Treatment of Patients With Connective Tissue Disease
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040077; 04-CH-0077
Record Dates: First submitted 2006-07-12; First posted 2004-02-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01-09

CONDITIONS: Connective Tissue Disorders; Osteogenesis Imperfecta; Bone Diseases, Metabolic; Melorheostosis
Keywords: Bone; Growth; Skin; Fractures
MeSH Terms: conditions — Connective Tissue Diseases; Osteogenesis Imperfecta; Bone Diseases, Metabolic; Melorheostosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled cohort: All patients enrolled, as this is an evaluation/diagnostic study

SUMMARY:
This study offers evaluation and treatment of patients with a suspected connective tissue disorder. The protocol is not designed to test new treatments; rather, patients receive standard care. The study is designed to: 1) allow NICHD's staff to learn more about connective tissue disorders, 2) train physicians in the evaluation and treatment of these disorders; and 3) establish a pool of patients who may be eligible for other NICHD protocols for connective tissue disorders. (Participants in this protocol will not be required to join another study; the decision will be voluntary.)

Patients of all ages with a suspected connective tissue disorder and their unaffected family members may be eligible for this study.

Participants undergo diagnostic procedures that may include a medical history, physical examination, X-ray studies, eye examinations, and blood drawing, as well as other specialized tests, when needed. Additional tests may include:

* Blood test for DNA genetic analysis
* Skin biopsy: Removal of a small piece of tissue for microscopic examination. The area of skin selected for the biopsy is numbed and a small circle of skin, usually from the upper arm, is removed with a surgical cookie cutter-like instrument.
* Magnetic resonance imaging (MRI): This test uses a strong magnetic field and radio waves to show structural and chemical changes in tissues. The patient lies on a table that slides into a narrow cylinder containing a magnetic field. Ear plugs are worn to muffle loud knocking and thumping sounds that occur with electrical switching of the magnetic fields.
* Computed tomography (CT) scans: This test allows the doctor to view the organs inside the body in small sections. The patient lies in a doughnut-like machine. Scanning can be done from different angles, allowing a three dimensional picture of the part of the body being studied. It may be done with or without injection of a contrast material.
* Referral to appropriate sub-specialists when potential complications are found.

DETAILED DESCRIPTION:
This protocol seeks to formalize the application of accepted diagnostic and therapeutic measures in the study of individuals with known or suspected bone-related connective tissue disorders, including Osteogenesis Imperfecta and melorheostosis. It is our intent to attract a broad array of such individuals for the purposes indicated above. This protocol will also serve as a basis for permitting collaborations with other investigators regarding rare, illustrative, or poorly defined human diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals with a suspected bone-related connective tissue disorder, as indicated by signs including, but not limited to, fractures, low bone density, asymmetric overgrowth of long bone

OR

Apparently unaffected, healthy family members of individuals with a suspected bone-related connective tissue disorder.

Ages to be enrolled are from 0-70 years old, with only viable neonates accepted at age 0 years.

EXCLUSION CRITERIA:

Individuals who, in the opinion of the Investigator, are unable to comply with the protocol or have medical conditions that would potentially increase the risk of participation.

For both affected individuals and apparently healthy family members, no exclusions are based on age, gender, ethnicity or race, religion, or English-language ability. Those who are pregnant, whether affected or unaffected, will be excluded from any exam that includes

radiation, but not excluded from the study overall.

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Minimal limit on gender, geographical location (able to travel to NIH), race/ethnicity, age (from birth to 70 years old).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2004-05-18 (Actual)

PRIMARY OUTCOMES:
Evaluation and Diagnosis | per individual cases
  Evaluation of individuals with suspected bone-related connective tissue disorders and their family members

SECONDARY OUTCOMES:
Biospecimens collection | 12/31/2030
  Collection of biospecimens for use in clinical and basic science research of bone-related connective tissue disorders and controls

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Zimmerberg, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The intention of this study is for individualized, very rare explorations of conditions that may lead to clearer diagnoses for patients and/or open up avenues of further study by qualification for other trials by providing diagnosis or clinical information relevant to that disease process such as osteogenesis imperfecta or melorheostosis studies. It also allows for family member analysis of these genetic conditions for those apparently unaffected. It is considered a screening study. The IPD will not be shared as a cohort, though individual plans will be made later for those whose case studies would be published directly from data received on this protocol.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-CH-0077.html